CLINICAL TRIAL: NCT06553729
Title: Effects of Vitamin D and Prebiotic Supplementation on Glucose Control During Pregnancy: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial
Brief Title: Effects of Vitamin D and Prebiotic Supplementation on Glucose Control During Pregnancy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, An Pan, Professor, Huazhong University of Science and Technology
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VD, Prebiotics in Pregnancy
Record Dates: First submitted 2024-08-11; First posted 2024-08-14 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Glucose Intolerance During Pregnancy
Keywords: Vitamin D; Prebiotics; Glucose Intolerance During Pregnancy; Blood Glucose; Gestation diabetes; Adverse pregnancy outcomes
MeSH Terms: interventions — Cholecalciferol; Prebiotics; Inulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Vitamin D3 + Prebiotics (Active Comparator): Vitamin D3 (cholecalciferol), 1600 IU per day. Prebiotics (inulin), 10g per day.
  Interventions: Drug: Vitamin D3; Dietary Supplement: Prebiotics
- Vitamin D3 + Prebiotics placebo (Active Comparator): Vitamin D3 (cholecalciferol), 1600 IU per day. Prebiotics placebo.
  Interventions: Drug: Vitamin D3; Dietary Supplement: Prebiotics placebo
- Prebiotics +Vitamin D3 placebo (Active Comparator): Prebiotics (inulin), 10g per day. Vitamin D3 placebo.
  Interventions: Dietary Supplement: Prebiotics; Dietary Supplement: Vitamin D3 placebo
- Vitamin D3 placebo + Prebiotics placebo (Placebo Comparator): Vitamin D3 placebo. Prebiotics placebo.
  Interventions: Dietary Supplement: Prebiotics placebo; Dietary Supplement: Vitamin D3 placebo

INTERVENTIONS:
Drug: Vitamin D3 — Vitamin D3 (cholecalciferol), 1600 IU per day.
  Other Names: Cholecalciferol
  Arms: Vitamin D3 + Prebiotics; Vitamin D3 + Prebiotics placebo
Dietary Supplement: Prebiotics — Prebiotics (inulin), 10g per day.
  Other Names: Inulin
  Arms: Prebiotics +Vitamin D3 placebo; Vitamin D3 + Prebiotics
Dietary Supplement: Prebiotics placebo — Prebiotics placebo.
  Arms: Vitamin D3 + Prebiotics placebo; Vitamin D3 placebo + Prebiotics placebo
Dietary Supplement: Vitamin D3 placebo — Vitamin D3 placebo
  Arms: Prebiotics +Vitamin D3 placebo; Vitamin D3 placebo + Prebiotics placebo

SUMMARY:
The goal of this randomized, double-blind, placebo-controlled study included pregnant women at high risk of GDM at 6-15 weeks of gestation is to investigate whether supplementation with vitamin D (1600 IU per day) or prebiotics (inulin, 10 gram per day) during pregnancy has beneficial effects on controlling blood glucose during pregnancy.

DETAILED DESCRIPTION:
The goal of this randomized, double-blind, placebo-controlled study included pregnant women at high risk of GDM at 6-15 weeks of gestation is to investigate whether supplementation with vitamin D (1600 IU per day) or prebiotics (inulin, 10 gram per day) during pregnancy has beneficial effects on controlling blood glucose during pregnancy.

About 500 pregnant women aged 18-45 years, at 6-15 weeks of gestation, had resided locally for at least one year, with high risk of GDM will be enrolled in the study. Pregnant women at high risk of GDM are defined as meeting any of the following criteria:

1. Pre-pregnancy body mass index (BMI) ≥24.0 kg/m2;
2. History of GDM or a family history of diabetes;
3. History of delivery of macrosomia (birth weight >4000 g);
4. Glycated hemoglobin (HbA1c) 5.7-6.4% or fasting blood glucose 5.6-7.0 mmol/L; Eligible participants must have singleton pregnancy, no infertility treatment, no history of diabetes or a definite diagnosis of diabetes, or impaired glucose tolerance at recruitment (fasting blood glucose >7.0 mmol/L or HbA1c≥6.5%), no allergic history of chicory root and they will be required to agree to limit the use of vitamin D, prebiotics, probiotics, or synbiotic supplementations and to be convenient access to study centers. Safety exclusions include serious chronic or infectious diseases, serious liver or kidney disease, abnormalities in calcium metabolism, and clinically diagnosed mental disorders, or other conditions that would preclude participation.

Eligible participants will be assigned by chance to one of four groups: (1) daily vitamin D (1600 IU) and prebiotics (10 gram); (2) daily vitamin D (1600 IU) and prebiotics placebo; (3) daily vitamin D placebo and prebiotics (10 gram); or (4) daily vitamin D placebo and prebiotics placebo. Randomization will be conducted.

At enrollment, baseline questionnaires are designed to collect data on sociodemographic factors, pregnancy-related information, lifestyle habits, health status, and medical conditions before and during pregnancy. Participants in all groups will take two capsules that contained either vitamin D or vitamin D placebo and a strip of prebiotics powder (10 g per strip, brew with warm water and take with meals) or prebiotics placebo each day until delivery.

Participants will be followed up three times during pregnancy (24-28 weeks gestation, 32-36 weeks gestation and delivery), and receive a single stage-specific dosage at any given follow-up time.

Participants will have physical measurements of height, weight, other anthropometric measurements, and blood pressure at baseline and each follow-up visit. Blood, urine, and stool samples will also be obtained in the study center, fasting blood glucose, HbA1c and other biochemical indicators will also be detected at the same time, and a 75g oral glucose tolerance test (OGTT) will be measured during 24-28 weeks of gestation to diagnose GDM.

The primary outcomes, including fasting blood glucose and HbA1c will be measured using blood samples.

Secondary outcomes in this study include incidence of GDM, changes in blood lipids (such as total cholesterol, triglycerides, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol), trends in plasma vitamin D levels, inflammatory factors, intestinal flora related indicators, delivery mode, incidence of preeclampsia and adverse pregnancy outcomes. Data will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. 6-15 weeks of gestation.
2. Age 18-45 years old.
3. Permanent resident or resident locally at least one year.
4. GDM high-risk pregnant women (meeting any of the following criteria):

   1. Pre-pregnancy body mass index (BMI) ≥24.0 kg/m2,
   2. History of GDM or a family history of diabetes,
   3. History of delivery of macrosomia (birth weight >4000 g),
   4. HbA1c 5.7-6.4% or fasting blood glucose 5.6-7.0 mmol/L.

Exclusion Criteria:

1. Multiple pregnancy.
2. Have received infertility treatment such as in vitro fertilization or intrauterine insemination.
3. History of diabetes or current diagnosis of diabetes (including type 1 and type 2 diabetes) or abnormal glucose tolerance at recruitment (fasting blood glucose >7.0 mmol/L or HbA1c≥6.5%).
4. Serious chronic diseases (including cardiovascular and cerebrovascular diseases, cancer, and thyroid dysfunction) or infectious diseases (including hepatitis B, active tuberculosis, acquired immunodeficiency syndrome, and syphilis).
5. Severe liver disease (such as cirrhosis) or severe kidney disease (such as renal failure or requiring dialysis).
6. Kidney stones, hypercalcemia, hypercalciuria, parathyroid hormone abnormality.
7. Any mental disorders, such as schizophrenia, depression, other mental disorders, or bipolar disorder.
8. History of allergy or intolerance to vitamin D, chicory root, or starch.
9. Have participated in or are participating in other clinical trials within the past 3 months.
10. Daily vitamin D intake >800 IU.
11. Inability or refusal to answer and communicate.
12. Those who are unwilling to sign the informed consent.
13. The researcher thinks that it is not suitable to participate in this research.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Concentration of fasting blood glucose | 24-28 gestational weeks, 32-36 gestational weeks, and delivery
  Concentration of fasting blood glucose, measured in mmol/L
Glycated hemoglobin (HbA1c) | 24-28 gestational weeks, 32-36 gestational weeks, and delivery
  Concentration of HbA1c, measured in the percentage of hemoglobin

SECONDARY OUTCOMES:
Incidence of Gestational Diabetes | 24-28 gestational weeks
  75g oral glucose tolerance test (OGTT) will be performed at 24-28 weeks of gestation to diagnose gestational diabetes
Concentration of blood lipids | 24-28 gestational weeks, 32-36 gestational weeks, and delivery
  Concentration of blood lipids (total cholesterol, triglycerides, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol), measured in mmol/L
Concentration of plasma 25(OH)D | 24-28 gestational weeks, 32-36 gestational weeks, and delivery
  Concentration of plasma 25(OH)D concentrations, measured in nmol/L
Concentration of C-reactive protein (CRP) | 24-28 gestational weeks, 32-36 gestational weeks, and delivery
  Concentration of CRP, measured in mg/dL
Concentration of interleukin-6 (IL-6) | 24-28 gestational weeks, 32-36 gestational weeks, and delivery
  Concentration of IL-6, measured in pg/mL
Metagenomic analysis of the gut microbiota | 24-28 gestational weeks, 32-36 gestational weeks, and delivery
  The diversity of the gut microbiota will be assessed by high-quality whole-metagenomic sequencing
Birth weight | Delivery
  The baby's weight at birth, Weight in grams
Gestational duration | Delivery
  The length of a woman's pregnancy from the start of her last period, duration in days
Delivery mode | Delivery
  Method of the baby being born during childbirth, vaginal delivery or cesarean section

CONTACTS AND LOCATIONS:
Overall Officials: Gang Liu, PHD, Principal Investigator — School of Public Health, Tongji Medical College, Huazhong University of Science and Technology; An Pan, PHD, Principal Investigator — School of Public Health, Tongji Medical College, Huazhong University of Science and Technology
Locations (2):
- China (2):
  - Central People's Hospital of Zhanjiang, Zhanjiang, Guangdong
  - Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei

IPD SHARING:
Plan to Share IPD: No